CLINICAL TRIAL: NCT01045668
Title: Comparison of the Effect of Ablation of the Clinically Presenting Ventricular Tachycardia (VT) Only Versus the Addition of Substrate Ablation Based on Scar Mapping; on the Long Term Success Rate of VT Ablation
Brief Title: Ablation of Clinical Ventricular Tachycardia Versus Addition of Substrate Ablation on the Long Term Success Rate of VT Ablation
Acronym: VISTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: University of Kansas (Other); California Pacific Medical Center (Other); Stanford University (Other); Case Western Reserve University (Other); Southlake Regional Health Centre (Other); Catholic University, Italy (Other); Ospedale dell'Angelo, Venezia-Mestre (Other); RCCS Monzino Hospital, Milan, Italy (Unknown); University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAI-VISTA
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical VT ablation (Active Comparator)
  Interventions: Procedure: Radiofrequency Catheter Ablation (RFCA)
- clinical VT and substrate ablation (Active Comparator)
  Interventions: Procedure: Radiofrequency Catheter Ablation (RFCA)

INTERVENTIONS:
Procedure: Radiofrequency Catheter Ablation (RFCA) — RFCA of clinical VT
  Arms: Clinical VT ablation
Procedure: Radiofrequency Catheter Ablation (RFCA) — RFCA of clinical VT as well as VT substrates
  Arms: clinical VT and substrate ablation

SUMMARY:
This study aims to assess whether a combined technique of substrate ablation and ablation of the clinically presenting VT at the site of early activation is superior to ablation of the clinically presenting VT alone, in enhancing long-term success of VT ablation.

DETAILED DESCRIPTION:
Background: VT is found mostly in patients with structural heart disease. It is classified using morphological criteria (monomorphic or polymorphic), duration of arrhythmia (sustained or non-sustained) or the mechanism of arrhythmia formation (re-entry, increased automation or triggered activity). The therapeutic approach and prognostic estimates of these different types of VT depend to a great degree on the mechanistic basis of the disease as well as the extent of myocardial damage and success of the therapy is measured by the absence of recurrence.

Myocardial infarction with subsequent induction of VT is observed as a consequence of coronary artery disease (CAD). The infarct regions that are morphologically and electrically diseased can be arrhythmogenic and may form the substrate for macro-reentrant VT.

Although antiarrhythmic drugs remain the primary form of therapy for VT, non-pharmacologic techniques like implantable cardioverter-defibrillator (ICD) and catheter ablation (CA) are becoming increasingly popular because of advancement in technology as well as an increase in desire among patients to eliminate the arrhythmia with ablation rather than suppressing it with drugs. ICDs and CA effectively terminate VT on a short-term basis; but multiple morphologies, hemodynamic instability and non-inducibility limit the long-term success rate of CA. The 'substrate mapping' approach defines areas of ventricular scar which can be potential VT sources. Several studies on small groups of patients have shown that successful ablation of VT substrates either reduces the recurrence of VT to 19- 50% or reduces the frequency of recurrence as well as the requirement of anti-arrhythmic drugs (AADs).

Study design:

This study is a multicenter, randomized, open label, parallel-arm clinical trial. A total of 120 post-myocardial infarction patients will be randomized at a 1:1 ratio into 2 groups:

1. ablation targeting the clinically presenting VT at the site of early activation only, or
2. ablation targeting the clinically presenting VT at the site of early activation plus substrate-based RF ablation

Follow-up:

Patients will undergo ICD interrogation at 3, 6 and 12 months to collect VT episode data, VT symptom assessment, complication assessment and AAD records. Management of AADs will be at the discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Previous Myocardial infarction
* Symptomatic, drug-refractory and haemodynamically stable VT following CAD
* Undergoing a VT ablation
* Implanted ICD

Exclusion Criteria:

* Documented valvular heart disease
* Acute myocardial infarction within the preceding 1 month
* Unstable angina
* Prolonged QT interval
* Patients with hemorrhagic or thrombophilic disorders
* Documented intra-atrial thrombus, tumor or other conditions which prevent easy catheter introduction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of any sustained VT in the post-ablation period as demonstrated by electronic documentation Procedural complications associated with prolonged use of radiofrequency (RF) energy such as perforation, cardiac tamponade | 48 hours

SECONDARY OUTCOMES:
Severe clinical events (hospital admissions for a cardiac cause, syncopal attacks, number of episodes of VT storms, death) Number of ICD interventions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD FACC FHRS, Principal Investigator — TCAI, St.David's Medical Center, Austin, TX
Locations (1):
- St.David's Medical Center, Austin, Texas, United States

REFERENCES:
- [Derived] Di Biase L, Burkhardt JD, Lakkireddy D, Carbucicchio C, Mohanty S, Mohanty P, Trivedi C, Santangeli P, Bai R, Forleo G, Horton R, Bailey S, Sanchez J, Al-Ahmad A, Hranitzky P, Gallinghouse GJ, Pelargonio G, Hongo RH, Beheiry S, Hao SC, Reddy M, Rossillo A, Themistoclakis S, Dello Russo A, Casella M, Tondo C, Natale A. Ablation of Stable VTs Versus Substrate Ablation in Ischemic Cardiomyopathy: The VISTA Randomized Multicenter Trial. J Am Coll Cardiol. 2015 Dec 29;66(25):2872-2882. doi: 10.1016/j.jacc.2015.10.026. PMID 26718674